CLINICAL TRIAL: NCT03686982
Title: The Impact of Supplementation With Novel Prototype Nutrition Bar on Nitric Oxide Bioavailability and Measures of Athlete Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1706
Record Dates: First submitted 2018-06-06; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Exercise Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Nitrate Bar (Experimental): include dietary nitrate; L-citrulline; epicatechin; vitamin C and glutathione
  Interventions: Other: Active Nitrate Bar
- Placebo Bar (Placebo Comparator): Containing no active ingredients
  Interventions: Other: Placebo Bar

INTERVENTIONS:
Other: Active Nitrate Bar — Bar containing Nitrate, L-citrulline; epicatechin; vitamin C and glutathione
  Arms: Active Nitrate Bar
Other: Placebo Bar — No active ingredients
  Arms: Placebo Bar

SUMMARY:
Dietary nitrate, L-citrulline, epicatechin, vitamin C and glutathione have the potential to improve nitric oxide (NO) bioavailability, in humans, by influencing both the nitrate-nitrite-NO and NO synthase-dependent pathways, and the storage of NO. The study is designed to assess the efficacy of a newly developed product containing a mixture of these compounds. Specifically, the study will assess if the product is capable of increasing NO bioavailability and if this results in positive effects on exercise economy and intermittent exercise performance. These outcome measures have been chosen because they have previously been positively impacted by an increase in NO bioavailability.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants in self-reported good general health as assessed by the standard procedures described below and specifically meeting the following blood pressure (BP) and body mass index (BMI) ranges: systolic BP: 100-140 mmHg; diastolic BP: 60-90 mmHg; and BMI 18.5-30.
2. 18-40 years of age
3. Physically active. Determined by meeting the following criteria: completes vigorous physical activity (i.e. activities that take hard physical effort and make you breathe much harder than normal; e.g. heavy lifting, digging, aerobics, fast cycling, running etc) at least 2 x per week and moderate physical activities (i.e. activities that take moderate physical effort and make you breath somewhat harder than normal; for example: carrying light loads, cycling at a regular pace, playing doubles tennis) at least 3 x per week.
4. Understanding of the procedures to be undertaken as part of the study
5. Willingness to participate in exercise testing and follow supplementation guidelines and other instructions provided by the experimenter
6. Informed, voluntary, written consent to participate in the study

Exclusion Criteria:

1. Known pulmonary, cardiovascular or metabolic disease
2. Food allergies including phenylketonurea (PKU)
3. Current regular use of any dietary supplement (excluding macronutrient based supplements) or previous use of any dietary supplement in the past 6 months that is known to have a lasting effect.
4. Blood donation within 3 months prior to the start of the study
5. Substance abuse within 2 years of the start of the study
6. Smoking
7. Any prescription and non-prescription medication which may impact saliva production (antidepressants, diuretics, analgesics, antihistamines, anti-hyper/hypo-tensives, anti-anxiety, appetite suppressants).
8. Current or previous use of phosphodiesterase 5 (PDE5) inhibitors.
9. Participation in another clinical trial within past 4 weeks.
10. Participation in another PepsiCo study within the past 6 months.
11. Highly trained or elite endurance athlete as determined by current or recent (within 3 months) participation in an endurance sport at international or national level.
12. Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Mean power output during intermittent exercise test | 5 days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andy Jones, PhD, Principal Investigator — University of Exeter, Sport and Health Sciences department
Locations (1):
- University of Exeter, Sport and Health Sciences department,, Exeter, United Kingdom